CLINICAL TRIAL: NCT05769140
Title: Measurement of Cardiopulmonary Variables in a Large Group of Healthy Subjects with Acute Exposure to High Altitude
Brief Title: Measurement of Cardiopulmonary Variables After Acute Exposure to High Altitude
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Skyway Monte Bianco (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCM 1229
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: High Altitude Effects
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As altitude increases, the availability of oxygen in the air decreases, and just to compensate for this lack, the body increases cardiac and respiratory work and changes blood pressure. But that is not all: at altitude the body's ability to use oxygen is also limited. Thus, there is on one hand less oxygen available, and on the other a lower capacity to use it. All this generates significant alterations at the cardiovascular level, to the point of running possible risks of heart attack, stroke and acute pulmonary edema, particularly for individuals already suffering from cardiovascular disease.

The availability of modern cable cars allows an increasingly large number of individuals, including sedentary people, elderly subjects, and cardiorespiratory patients, to easily and rapidly reach high-altitude locations. Data on what happens on the cardiovascular system at high altitude are relatively scarce, and most experiments in the literature are limited by low sample sizes.

The primary purpose of this study is to assess the characteristics of a large population that acutely reached high altitude at Punta Helbronner (3,466 m above sea level), a location on Mont Blanc that is readily accessible by a 20-minute cableway ride from Courmayeur (Entreves station, 1,300 m, Skyway Monte Bianco). We aim to create a unique database and study correlations between altitude and cardiorespiratory parameters (heart rate, blood pressure, and Hb saturation) by collecting medical history data and biometric measurements in a very large population and to identify subjects most at risk of developing hypoxia at altitude. In a subset of subjects, differences in biometric variables after acute exposure at high altitude (in the transition between the downstream and the upstream measuring station) will be evaluated.

Two biometric multiparametric recording systems (Keito K9; Keito, Barcelona, Spain) were installed at Entreves station as well as at Punta Helbronner. Keito K9 is an automatic multiparametric recoding system for measuring peripheral oxygen saturation SpO2, heart rate HR (pulse oximeter), blood pressure (BP; wrist pressure cuff, automatic), height (laser height meter), weight (scale platform), and body mass index (BMI). Once initiated by the subject with the completion of a cardiology history questionnaire (self-reported), the automated Keito K9 system provides a sequence of vocal and animated directions to guide subjects through the measurements (the subject may elect to abstain from some of the measurements). Upon completion, the system prints a summary receipt for the subject, and the measurements are transmitted through a Wi-Fi network and collected in an Excel sheet.

It should be noted that all data collected will be anonymized or not traceable to the subject, through the use of a disposable identification card (for subjects who will perform both downstream and upstream measurement).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive volunteer subjects accessing the Skyway Monte Bianco cableway and stopping to take measurements at the two biometric multiparametric recording systems Keito K9
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
relationship between oxygen saturation after acute exposure to high altitude and age | immediately after the evaluation
  determine if there is a relationship between oxygen saturation as % (pulse oximeter included in the biometric station) and age (self-reported in automated questionnaire included in the biometric station software and created ad hoc by research team) following acute exposure to high altitude
relationship between oxygen saturation after acute exposure to high altitude and sex | immediately after the evaluation
  determine if there is a relationship between oxygen saturationas % (pulse oximeter included in the biometric station) and sex (self-reported in automated questionnaire included in the biometric station software and created ad hoc by research team) following acute exposure to high altitude
relationship between oxygen saturation after acute exposure to high altitude and heart rate | immediately after the evaluation
  determine if there is a relationship between oxygen saturation % (pulse oximeter included in the biometric station) and heart rate (pulse oximeter included in the biometric station) following acute exposure to high altitude
relationship between oxygen saturation after acute exposure to high altitude and blood pressure | immediately after the evaluation
  determine if there is a relationship between oxygen saturation (pulse oximeter included in the biometric station) and blood pressure (automatic wrist pressure cuff included in the biometric station) following acute exposure to high altitude
relationship between oxygen saturation after acute exposure to high altitude and BMI | immediately after the evaluation
  determine if there is a relationship between oxygen saturation (pulse oximeter included in the biometric station) and body mass index (calculated from height (laser height meter) and weight (scale platform)) following acute exposure to high altitude

SECONDARY OUTCOMES:
study the delta of oxygen saturation introduced by acute exposure to high altitude | immediately after the evaluation
  study the delta of oxygen saturation (pulse oximeter) introduced by acute exposure to high altitude (differences in this variable in the transition between the downstream and the upstream measuring station)
study the delta of heart rate introduced by acute exposure to high altitude | immediately after the evaluation
  study the delta of heart rate (pulse oximeter) introduced by acute exposure to high altitude (differences in this variable in the transition between the downstream and the upstream measuring station)
study the delta of blood pressure introduced by acute exposure to high altitude | immediately after the evaluation
  study the delta of blood pressure (automatic wrist pressure cuff) introduced by acute exposure to high altitude (differences in this variable in the transition between the downstream and the upstream measuring station)

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, Prof, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Skyway Monte Bianco, Courmayeur, Aosta, Italy

IPD SHARING:
Plan to Share IPD: No